CLINICAL TRIAL: NCT01928290
Title: Phase II Study of FOLFIRINOX Chemotherapy for Treatment of Advanced Gastric, Gastro-esophageal Junction, and Esophageal Tumors
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Stomach, Gastroesophageal, or Esophageal Cancer
Acronym: FOLFIRINOX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201309035
Record Dates: First submitted 2013-08-19; First posted 2013-08-23 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Stomach Neoplasms; Esophageal Neoplasms
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms | interventions — Irinotecan; Trastuzumab; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: FOLFIRINOX (HER2-negative) (Experimental): Irinotecan 180 mg/m2 IV on Days 1 & 15.
  Oxaliplatin 85 mg/m2 IV on Days 1 & 15.
  Leucovorin 400 mg/m2 IV on Days 1 & 15.
  Fluorouracil 400 mg/m2 bolus and 2400 mg/m2 CIVI over 46 hours beginning on Day 1 and Day 15.
  Interventions: Drug: Irinotecan; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil
- Arm B: FOLFIRINOX & Trastuzumab (HER2-positive) (Experimental): Trastuzumab 8 mg/kg on Cycle 1 Day 1 then 4 mg/kg on Day 15 and Day 1 of all future cycles.
  Irinotecan 180 mg/m2 IV on Days 1 & 15.
  Oxaliplatin 85 mg/m2 IV on Days 1 & 15.
  Leucovorin 400 mg/m2 IV on Days 1 & 15.
  Fluorouracil 400 mg/m2 bolus and 2400 mg/m2 CIVI over 46 hours beginning on Day 1 and Day 15.
  Interventions: Drug: Irinotecan; Drug: Trastuzumab; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil

INTERVENTIONS:
Drug: Irinotecan
  Other Names: Camptosar®; CPT-11
Drug: Trastuzumab
  Other Names: Herceptin®
  Arms: Arm B: FOLFIRINOX & Trastuzumab (HER2-positive)
Drug: Oxaliplatin
  Other Names: Eloxatin®
Drug: Leucovorin
  Other Names: Wellcovorin® I.V.; citrovorum factor
Drug: Fluorouracil
  Other Names: folinic acid; 5-formyl tetrahydrofolate; Adrucil® Injection; 5-Fluorouracil; 5-FU

SUMMARY:
This phase II trial studies how well combination chemotherapy works in treating patients with advanced stomach, gastroesophageal, or esophageal cancer. Drugs used in chemotherapy, such as irinotecan hydrochloride, oxaliplatin, leucovorin calcium, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven and inoperable locally advanced, recurrent, or metastatic cancer of the esophagus, stomach, or gastro-esophageal junction.
2. Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥10 mm with CT scan, as ≥20 mm by chest x-ray, or ≥10 mm with calipers by clinical exam.
3. Prior single modality radiation therapy is allowed.
4. At least 18 years of age.
5. ECOG performance status ≤ 2
6. Normal bone marrow and organ function as defined below:

   1. Absolute neutrophil count ≥ 1,500/mcl
   2. Platelets ≥ 100,000/mcl
   3. AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN
   4. Creatinine ≤ IULN OR creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
   5. LVEF ≥ 50%
7. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
8. Ability to understand and willingness to sign an IRB approved written informed consent document (legally authorized representative is allowed).
9. Patients already receiving treatment with FOLFIRINOX +/- trastuzumab may participate in the study and have their data collected retrospectively if they met inclusion criteria at the start of therapy and sign consent for study participation moving forward.

Exclusion Criteria:

1. Chemotherapy in the 6 months prior to registration.
2. Any active malignancy within 3 years that may alter the course of esophageal cancer (Apparently cured localized malignancy or advanced, but indolent malignancy with significantly more favorable prognosis are allowed)
3. Receiving any other investigational agents at the time of registration.
4. Known untreated brain metastases. These patients must be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
5. A history of allergic reactions attributed to compounds of similar chemical or biologic composition to the agents used in the study.
6. Previous therapy for metastatic gastroesophageal cancer. Previous perioperative chemotherapy is allowed as long as the duration without treatment has been greater than 6 months..
7. A history of congestive heart failure, transmural myocardial infarction, symptomatic valvular disease, or high-risk arrhythmia.
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
9. Pregnant and/or breastfeeding. Patient must have a negative urine pregnancy test within 14 days of study entry.
10. Known HIV-positivity and on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with trastuzumab. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Inclusion of Women and Minorities

Both men and women and members of all races and ethnic groups are eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-11-08 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2019-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haeseong Park, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park H, Jin RU, Wang-Gillam A, Suresh R, Rigden C, Amin M, Tan BR, Pedersen KS, Lim KH, Trikalinos NA, Acharya A, Copsey ML, Navo KA, Morton AE, Gao F, Lockhart AC. FOLFIRINOX for the Treatment of Advanced Gastroesophageal Cancers: A Phase 2 Nonrandomized Clinical Trial. JAMA Oncol. 2020 Aug 1;6(8):1231-1240. doi: 10.1001/jamaoncol.2020.2020. PMID 32469386
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 11/08/2013 and closed to participant enrollment on 07/23/2018.
Period: Overall Study
Arm/Group | Arm A: FOLFIRINOX (HER2-negative) | Arm B: FOLFIRINOX & Trastuzumab (HER2-positive)
Started | 41 | 26
Completed | 41 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: FOLFIRINOX (HER2-negative) | Arm B: FOLFIRINOX & Trastuzumab (HER2-positive) | Total
Number analyzed (Participants) | 41 | 26 | 67
Age, Continuous [Median (Full Range); unit: years] | 59 [43 to 78] | 59.5 [34 to 73] | 59 [34 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 0 | 11
  Male | 30 | 26 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 41 | 26 | 67
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 38 | 25 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 41 | 26 | 67

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Objective Response
Description: * Objective response (defined as complete response (CR) + partial response (PR) by RECIST 1.1 criteria)
  * CR: Disappearance of all target lesions, non-target lesions, and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Through completion of treatment (estimated to be 4 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: FOLFIRINOX (HER2-negative) | Arm B: FOLFIRINOX & Trastuzumab (HER2-positive)
Number analyzed (Participants) | 41 | 26
Participants | 25 | 22

2. Secondary Outcome: Progression Free Survival
Description: Duration of time from start of treatment to time of progression or death, whichever occurs first.
Time Frame: Through 1 year after completion of treatment (median follow-up 16.2 months - 95% CI 4.7-42.5 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: FOLFIRINOX (HER2-negative) | Arm B: FOLFIRINOX & Trastuzumab (HER2-positive)
Number analyzed (Participants) | 41 | 26
months | 8.4 [6.8 to 12.2] | 13.8 [10.0 to 19.8]

3. Secondary Outcome: Time to Progression (TTP)
Description: Duration of time from start of treatment to time of progression. Progression is defined as At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Through 1 year after completion of treatment (median follow-up 16.2 months - 95% CI 4.7-42.5 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: FOLFIRINOX (HER2-negative) | Arm B: FOLFIRINOX & Trastuzumab (HER2-positive)
Number analyzed (Participants) | 41 | 26
months | 8.0 [6.7 to 12.0] | 13.9 [9.9 to 19.5]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time interval from date of diagnosis to date of death from any cause.
Time Frame: Through 1 year after completion of treatment (median follow-up 16.2 months - 95% CI 4.7-42.5 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: FOLFIRINOX (HER2-negative) | Arm B: FOLFIRINOX & Trastuzumab (HER2-positive)
Number analyzed (Participants) | 41 | 26
months | 15.5 [10.6 to 19.6] | 19.6 [16.1 to 24.6]

5. Secondary Outcome: Clinical Benefit Rate
Description: * Clinical benefit rate is the percentage of combined patients who have achieved complete response (CR), partial response (PR), and stable disease (SD)
  * CR: Disappearance of all target lesions, non-target lesions, and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm
  * PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters
  * SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Through completion of treatment (estimated to be 4 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: FOLFIRINOX (HER2-negative) | Arm B: FOLFIRINOX & Trastuzumab (HER2-positive)
Number analyzed (Participants) | 41 | 26
Participants | 33 | 22

6. Secondary Outcome: Duration of Response
Description: Time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented
Time Frame: Through 1 year after completion of treatment (median follow-up 16.2 months - 95% CI 4.7-42.5 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: FOLFIRINOX (HER2-negative) | Arm B: FOLFIRINOX & Trastuzumab (HER2-positive)
Number analyzed (Participants) | 25 | 22
months | 5.8 [3.5 to 13.5] | 10.5 [7.9 to 18.4]

7. Secondary Outcome: Toxicity and Tolerability (Arm A and Arm B) as Measured by the Number of Participants With Grade 3 or Higher Adverse Events
Time Frame: 30 days after completion of treatment (estimated to be 5 months)
Measure: Number; unit: participants
Arm/Group | Arm A: FOLFIRINOX (HER2-negative) | Arm B: FOLFIRINOX & Trastuzumab (HER2-positive)
Number analyzed (Participants) | 41 | 26
participants
  Anemia | 1 | 0
  Febrile neutropenia | 2 | 0
  Anal Fistula | 1 | 0
  Diarrhea | 4 | 5
  Hematemesis | 1 | 0
  Nausea | 2 | 2
  Peripheral ischemia | 1 | 0
  Vomiting | 3 | 1
  Fatigue | 4 | 0
  Laparoscopy surgery | 1 | 0
  Pain | 1 | 0
  Sepsis | 1 | 0
  Lung infection | 1 | 0
  Pneumonia | 1 | 0
  Hypernatremia | 1 | 0
  Neutrophil count decreased | 19 | 8
  Platelet count decreased | 3 | 0
  Anorexia | 3 | 0
  Dehydration | 4 | 0
  Hypokalemia | 1 | 2
  Back pain | 1 | 0
  Peripheral sensory neuropathy | 2 | 0
  Syncope | 1 | 1
  Dyspnea | 1 | 0
  Pleural embolism | 1 | 0
  Skin infection | 1 | 0
  Thromboembolic event | 4 | 0
  Abdominal pain | 0 | 1
  Enterocolitis | 0 | 1
  Hemorrhoids | 0 | 1
  G-tube infection | 0 | 1
  Neutropenic entercolitis | 0 | 1
  Alkaline phosphatase increased | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment through 30 days following the last day of study treatment (up to 4 cycles following disease maximal response). All-cause mortality was collected through end of participant follow-up.
Description: For purposes of this study, abnormal lab values will only be collected and documented if they are clinically significant. Once a patient begins maintenance therapy, adverse events will no longer be collected and documented.
Arm/Group | Arm A: FOLFIRINOX (HER2-negative) | Arm B: FOLFIRINOX & Trastuzumab (HER2-positive)
All-Cause Mortality (participants affected / at risk) | 32/41 | 20/26
Serious Adverse Events (participants affected / at risk) | 18/41 | 8/26
Other Adverse Events (participants affected / at risk) | 41/41 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: FOLFIRINOX (HER2-negative) (N=41) | Arm B: FOLFIRINOX & Trastuzumab (HER2-positive) (N=26)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Death due to disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Edema limbs (General disorders) | 0 | 1
Enterocolitis (Infections and infestations) | 0 | 1
Fatigue (General disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Fever (General disorders) | 1 | 1
G-Tube infection (Infections and infestations) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Laparoscopy (Surgical and medical procedures) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 1
Neutropenic Enterocolitis (Gastrointestinal disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Peripheral ischemia (Gastrointestinal disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Vascular disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Thromboembolic event (Vascular disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: FOLFIRINOX (HER2-negative) (N=41) | Arm B: FOLFIRINOX & Trastuzumab (HER2-positive) (N=26)
Abdominal cramping (Gastrointestinal disorders) | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 11 | 5
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Agitation (Nervous system disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Alkaline phosphatase increased (Investigations) | 0 | 1
Allergic reaction (Immune system disorders) | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 20 | 6
Amnesia (Nervous system disorders) | 1 | 0
Anal Fistula (Gastrointestinal disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 3 | 1
Anorexia (Metabolism and nutrition disorders) | 19 | 6
Anxiety (Psychiatric disorders) | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Bladder pain (Renal and urinary disorders) | 1 | 0
Bloating (Gastrointestinal disorders) | 2 | 4
Blood bilirubin increased (Investigations) | 1 | 0
Blood in stool (Gastrointestinal disorders) | 1 | 0
Blurred vision (Eye disorders) | 5 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Brittle nails (Skin and subcutaneous tissue disorders) | 2 | 0
Bruising (Injury, poisoning and procedural complications) | 4 | 2
Catheter related infection (Infections and infestations) | 0 | 1
Chest tightening (Blood and lymphatic system disorders) | 0 | 1
Chills (General disorders) | 2 | 6
Cold sores on the nose (Skin and subcutaneous tissue disorders) | 1 | 0
Cold symptoms (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 16 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Crack in fingernails (Skin and subcutaneous tissue disorders) | 0 | 1
Cramping (Musculoskeletal and connective tissue disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Depression (Psychiatric disorders) | 7 | 2
Diarrhea (Gastrointestinal disorders) | 25 | 12
Dizziness (Nervous system disorders) | 13 | 3
Double vision (Eye disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0
Dysgeusia (Nervous system disorders) | 5 | 5
Dyspepsia (Gastrointestinal disorders) | 5 | 1
Dysphagia (Gastrointestinal disorders) | 4 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Dyspnea atrial fibrillation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Edema limbs (General disorders) | 9 | 2
Edema trunk (General disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 2
Esophageal pain (Gastrointestinal disorders) | 1 | 0
Esophageal stenosis (Gastrointestinal disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fatigue (General disorders) | 20 | 9
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Fever (General disorders) | 2 | 2
Flatulence (Gastrointestinal disorders) | 11 | 2
Floaters (Eye disorders) | 1 | 0
Flu Like Symptoms (General disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 0
Foot drop (Musculoskeletal and connective tissue disorders) | 0 | 1
GERD (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 10 | 2
Hearing imparied (Ear and labyrinth disorders) | 1 | 0
Hematemesis (Gastrointestinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Hoarseness (Gastrointestinal disorders) | 1 | 0
Hot flashes (Vascular disorders) | 4 | 2
Hypernatremia (Investigations) | 1 | 0
Hypertension (Vascular disorders) | 2 | 2
Hypokalemia (Metabolism and nutrition disorders) | 3 | 2
Infection near port (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (General disorders) | 4 | 0
Insomnia (Psychiatric disorders) | 4 | 5
Irritability (General disorders) | 1 | 0
Jaw pain (General disorders) | 0 | 1
Jittery (Psychiatric disorders) | 1 | 1
Laryngeal infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Leg cramping (Musculoskeletal and connective tissue disorders) | 1 | 0
Leg cramps (General disorders) | 0 | 1
Lost vision (Eye disorders) | 1 | 0
Lower heartrate (Cardiac disorders) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 13 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 20 | 8
Neutrophil count decreased (Investigations) | 19 | 8
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 2 | 0
Pain (General disorders) | 2 | 0
Pain around port (General disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Painful deep breaths (General disorders) | 1 | 0
Palmar Plantar Erythrodysesthia Syndrome (Skin and subcutaneous tissue disorders) | 3 | 0
Papulopustular rash (Skin and subcutaneous tissue disorders) | 2 | 0
Paresthesia (Nervous system disorders) | 3 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 26 | 11
Platelet count decreased (Investigations) | 5 | 0
Pleural embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 | 0
Rash maculo popular (Skin and subcutaneous tissue disorders) | 2 | 2
Rash on face (Skin and subcutaneous tissue disorders) | 0 | 1
Rash on forearms and neck (Skin and subcutaneous tissue disorders) | 0 | 1
Rectal pain (Gastrointestinal disorders) | 0 | 1
Rigors (General disorders) | 0 | 1
Runny nose (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sensitive nose (General disorders) | 1 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Sinus (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sore tongue (General disorders) | 1 | 0
Spasticity (Nervous system disorders) | 0 | 1
Superficial thrombophlebitis (Vascular disorders) | 0 | 1
Sweating (Skin and subcutaneous tissue disorders) | 1 | 2
Sweating after eating (Skin and subcutaneous tissue disorders) | 1 | 0
Swollen glands (General disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Tender gums (Gastrointestinal disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 4 | 2
Toothache (Gastrointestinal disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Upper respiratory infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Vaginal infection (Reproductive system and breast disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 13 | 3
Watering eyes (Eye disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT01928290/Prot_SAP_000.pdf